CLINICAL TRIAL: NCT00765973
Title: A Phase 1 Study of Topotecan Liposomes Injection (TLI) in Subjects With Small Cell Lung Cancer (SCLC), Ovarian Cancer and Other Advanced Solid Tumors
Brief Title: Topotecan Liposomes Injection for Small Cell Lung Cancer (SCLC), Ovarian Cancer and Other Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBS601
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Small Cell Lung Cancer; Ovarian Cancer; Solid Tumors
Keywords: Other Advanced Solid Tumors
MeSH Terms: conditions — Small Cell Lung Carcinoma; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Arm A: TLI dose on Days 1 and 8 of a 21-day treatment cycle (Starting dose: 1 mg/m2)
  Interventions: Drug: Topotecan Liposomes Injection (TLI)
- B (Experimental): Arm B: TLI dose on Day 1 of a 21-day treatment cycle (Starting dose: 2 mg/m2)
  Interventions: Drug: Topotecan Liposomes Injection (TLI)

INTERVENTIONS:
Drug: Topotecan Liposomes Injection (TLI) — TLI dose on Days 1 and 8 of a 21-day treatment cycle (Starting dose: 1 mg/m2)
  Arms: A
Drug: Topotecan Liposomes Injection (TLI) — TLI dose on Day 1 of a 21-day treatment cycle (Starting dose: 2 mg/m2)
  Arms: B

SUMMARY:
A multi-center, open-label, two-arm, dose-escalation study to establish the safety, tolerability, MTD, and schedule of TLI administered intravenously as a 30 minute infusion in adult subjects with advanced solid tumors that have relapsed, are refractory to standard therapy, or for whom there is no standard therapy available.

The two dosing regimens to be evaluated are:

* Arm A: TLI dose on Days 1 and 8 of a 21-day treatment cycle (Starting dose: 1 mg/m2)
* Arm B: TLI dose on Day 1 of a 21-day treatment cycle (Starting dose: 2 mg/m2)

When one of the two arms reaches MTD, all future subjects will then be enrolled in the remaining study arm until MTD of that arm is reached.

DETAILED DESCRIPTION:
The study will utilize an accelerated design with small initial cohort sizes that allow fewer subjects to be enrolled at sub-therapeutic doses such as the very low starting doses in both arms of the study. Initial cohorts will include only one subject and dose escalations will be in 100% increments until a single Grade 2 toxicity related to study drug or DLT occurs in Cycle 1. Dose escalation will proceed until the MTD is exceeded. MTD is defined as average of the highest dose level for which 2 out of 6 subjects experience a DLT and the previous dose level, provided no additional DLTs occur. Subjects who discontinue TLI treatment before completion of Cycle 1 for reasons other than toxicity will not be evaluable for the determination of MTD and will be replaced.

The study will consist of a screening period, treatment period, and a post-treatment period. Subjects will be followed for 30 days after their last TLI dose. Safety and tolerability parameters include clinical laboratory assessments, vital signs, physical examinations, and adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologically or cytologically confirmed advanced solid tumor that has relapsed, is refractory to standard treatment, or for whom there is no standard therapy available.
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
4. Normal organ and marrow function as defined below within 14 days of study entry

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   2. Platelet count ≥100 x 109/L
   3. Hemoglobin ≥ 9 g/dL
   4. Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN), or 5 x ULN for subjects with liver metastases
   6. Serum creatinine ≤ 1.5 x ULN or calculated estimated creatinine clearance ≥ 50 mL/min/1.73m2 for subjects with creatinine levels above institutional normal based on the Cockcroft and Gault formula.
5. Never received prior TLI or topotecan HCl (Hycamtin®)
6. At least 4 weeks must have elapsed from the last dose of chemotherapy.
7. Life expectancy ≥ 3 months
8. Women of childbearing potential must have a negative urine or blood pregnancy test within 7 days prior to initiation of treatment.
9. If female, subject is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (e.g., hormonal contraceptive, intra-uterine device (IUD), diaphragm with spermicide, condom with spermicide or abstinence) from the screening visit through the duration of study participation.
10. If male, subject agrees to use an acceptable barrier method for contraception from the screening visit though the duration of study participation.
11. Before enrollment, the subject is capable of understanding and complying with parameters as outlined in the protocol and able to sign a written informed consent according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

1. Use of any investigational drugs, biologics, or devices within 28 days prior to study treatment or planned use during the course of the study.
2. Primary tumors of central nervous system (CNS). Symptomatic brain metastases (unless subject is stable without requirement of steroids and/or antiseizure medications for at least three months) or leptomeningeal tumor involvement. Imaging studies are not required to rule this out unless there is a clinical suspicion of CNS disease.
3. Prior chemotherapy or radiotherapy within 4 weeks of Day 1 of study (6 weeks for nitrosureas or mitomycin C).
4. Planned concurrent systemic therapy (cytotoxic and/or cytostatic) and/or radiotherapy during study treatment.
5. Less than 4 weeks have elapsed from the time of major surgery.
6. Subjects with a history of allergic reactions or sensitivity attributed to compounds of similar chemical or biologic composition to TLI, including known allergies to the ingredients comprising the liposome (e.g., cholesterol and/or sphingomyelin), which in the Investigator's opinion may put the subject at risk for significant reaction to the study drug.
7. Subjects who are pregnant or lactating.
8. Subjects known to be positive for human immunodeficiency virus (HIV), hepatitis C antibody, or hepatitis B surface antigen.
9. Prophylactic hematologic growth factors administered ≤ 2 weeks prior to start of treatment with TLI (excluding darbepoetin alfa and epoetin alfa).
10. Active infection or any serious underlying medical condition, which would impair the ability of the subject to receive protocol treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11-10 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety, tolerability and maximum tolerated dose of 2 different dosing schedules of TLI administered intravenously | 21 days following initial dose

SECONDARY OUTCOMES:
Assess the pharmacokinetic profile of TLI | 21 Day Cycle

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas